CLINICAL TRIAL: NCT00654602
Title: A 48 Week, Open Label, Non-Comparative, Multicentre, Phase IIIb Study to Evaluate the Efficacy and Safety of the Lipid-Regulating Agent Rosuvastatin in the Treatment of Subjects With Fredrickson Type IIa and Type IIb Dyslipidaemia, Including Heterozygous Familial Hypercholesterolaemia.
Brief Title: 48-wk Open Label Phase IIIb to Evaluate Efficacy and Safety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4522IL/0091; D3560C00091
Record Dates: First submitted 2008-04-03; First posted 2008-04-08 (Estimated); Last update posted 2009-05-28 (Estimated); Status verified 2009-05

CONDITIONS: Dyslipidaemia
Keywords: cholesterol; low density lipoproteins; dyslipidaemia; Rosuvastatin; Crestor
MeSH Terms: conditions — Dyslipidemias | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor
Behavioral: Maintenance of specific diet

SUMMARY:
The purpose of this study is to assess the efficacy and safety of rosuvastatin in reducing low density lipoprotein cholesterol levels to internationally recognised goals in subjects with dyslipidaemia.

ELIGIBILITY:
Inclusion Criteria:

* Fasting low density lipoprotein level as defined by the protocol.
* Fasting triglyceride level as defined by the protocol.

Exclusion Criteria:

* The use of lipid lowering drugs or dietary supplements after Visit 1.
* Active arterial disease eg Unstable angina, or recent arterial surgery.
* Blood lipid levels above the limits defined in the protocol.
* Uncontrolled hypertension, hypothyroidism, alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2002-02; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Reduction in low density lipoprotein cholesterol levels | 12 weeks

SECONDARY OUTCOMES:
Reduction in low density lipoprotein cholesterol levels | 24 & 48 weeks
Safety: adverse events & abnormal laboratory markers | 4 weekly until week 12 then 12 weekly thereafter.
Maintenance of lowered low density lipoprotein cholesterol level | Between week 12-48

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Evan Stein, Principal Investigator — Metabolic & Athersclerotic research centre, USA; Russell Esterline, Study Director — AstraZeneca